CLINICAL TRIAL: NCT06118463
Title: Study on AUNIP as a Novel Tumor Marker for Cervical Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Lin Yuan (Other)
Responsible Party: Sponsor-Investigator, Lin Yuan, Principal Investigator, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: yl20231001
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: Women aged 20-60; There is a definite pathological diagnosis of cervical cancer
  Interventions: Diagnostic Test: Detection of serum AUNIP expression
- Healthy control group: Women aged 20-60; No tumors in the uterus or other parts of the body; No inflammatory disease; Blood routine and blood biochemical tests are normal.
  Interventions: Diagnostic Test: Detection of serum AUNIP expression

INTERVENTIONS:
Diagnostic Test: Detection of serum AUNIP expression — The experiment is carried out according to the ELISA kit instructions, and the absorbance optic density (OD) value of the enzyme labeler at 450 nm is read. The protein concentration of AUNIP in the serum sample is calculated according to the standard curve.

SUMMARY:
To detect the expression of AUNIP in cervical cancer serum, and to clarify its diagnostic and prognostic value.

DETAILED DESCRIPTION:
Blood of all study participants of cervical cancer patients are collected to detect the expression of AUNIP, analyze the statistical correlation between the expression of cervical cancer AUNIP and clinicopathological parameters of patients, and preliminarily understand the expression of AUNIP in cervical cancer tumor tissues and its clinical diagnostic and progniostic value.

ELIGIBILITY:
Inclusion Criteria:

Study group inclusion criteria:

* Women aged 20-60
* There is a definite pathological diagnosis of cervical cancer

Healthy control group:

* Women aged 20-60
* No tumors in the uterus or other parts of the body
* No inflammatory disease
* Blood routine and blood biochemical tests are normal

Exclusion Criteria:

Exclusion criteria of the study group:

* There are other lesions in the uterus and uterine adnexa

Exclusion criteria of healthy control group:

* Pregnant, lactating or menarche women
* Women who are undergoing human papillomavirus (HPV) vaccination

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this study, 150 patients with cervical cancer in the First Affiliated Hospital of Shandong First Medical University (Shandong Qianfoshan Hospital) are selected as the study group. 150 healthy women are taken as control group during the same period.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
AUNIP expression in serum | through study completion, an average of 3 year
  Serum AUNIP expression is detected by ELISA kit. The results will be recorded seperately.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yuan, Ph.D., Principal Investigator — Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The plan will be shared after the clinial trial is completed and the patent protection is obtained.

REFERENCES:
- [Background] Yang Z, Liang X, Fu Y, Liu Y, Zheng L, Liu F, Li T, Yin X, Qiao X, Xu X. Identification of AUNIP as a candidate diagnostic and prognostic biomarker for oral squamous cell carcinoma. EBioMedicine. 2019 Sep;47:44-57. doi: 10.1016/j.ebiom.2019.08.013. Epub 2019 Aug 10. PMID 31409573
- [Background] Ma C, Kang W, Yu L, Yang Z, Ding T. AUNIP Expression Is Correlated With Immune Infiltration and Is a Candidate Diagnostic and Prognostic Biomarker for Hepatocellular Carcinoma and Lung Adenocarcinoma. Front Oncol. 2020 Dec 9;10:590006. doi: 10.3389/fonc.2020.590006. eCollection 2020. PMID 33363020